CLINICAL TRIAL: NCT05110937
Title: Dysfunctional Myelopoiesis and Myeloid-Derived Suppressor Cells in Sepsis Pathobiology Subtitle: Pathological Myeloid Activation After Sepsis and Trauma
Brief Title: Dysfunctional Myelopoiesis and Myeloid-Derived Suppressor Cells in Sepsis
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB202100559; RM1GM139690 (NIH); R35GM140806 (NIH)
Record Dates: First submitted 2021-10-14; First posted 2021-11-08 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Sepsis; Trauma Injury
MeSH Terms: conditions — Sepsis; Accidental Injuries | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sepsis: Blood collection: Blood will be collected from patient at day 4, day 7, day 14-21 and at 3 and 6 months.
  Interventions: Other: Blood sampling
- Healthy Controls: Blood Collection.
  The healthy volunteer participants will donate a blood sample. These controls will allow the investigators to determine if the values obtained are accurate, reliable, and repeatable.
  Interventions: Other: Blood sampling
- Trauma: Blood collection: Blood will be collected from patient at day 4, day 7, day 14-21 and at 3 and 6 months.
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Blood sampling

SUMMARY:
Adverse outcomes in surgical sepsis patients are secondary to dysregulated emergency myelopoiesis, and expansion of myeloid-derived suppressor cells. Here we propose to determine the underlying mechanisms behind the increased expansion of these leukocyte populations and the underlying mechanisms that drive inflammation and immune suppression.

DETAILED DESCRIPTION:
Our overarching hypothesis is that the consequences of surgical sepsis (death and poor quality of life) are the result of an unresolving host leukocyte dyscrasia, similar to other chronic conditions such as cancer and autoimmune disease. Specifically, the preferential expansion and self-perpetuation of myeloid-derived suppressor cells (MDSCs), propagated in part through epigenetic changes in both bone marrow (BM) progenitors and MDSCs, drives non-acute infectious and noninfectious complications after sepsis.

This Program will investigate in human surgical sepsis the underlying mechanisms that drive 'dysfunctional myelopoiesis', expansion of MDSC populations, suppressed T-cell quantities/function, and the development of patient's immunosuppressive/inflammatory endotypes. We will primarily focus on how MDSC expansion evolves over time in an observational study that follows surgical sepsis patients who do or do not rapidly recover. There are three specific aims: Aim 1. To test the hypothesis that perpetuation of host MDSCs after acute surgical sepsis drives poor long-term clinical outcomes in surgical sepsis, including but not limited to increased secondary infections. Aim 2. To test the hypothesis that failure to recover from surgical sepsis is driven by modifiable epigenetic alterations in circulating MDSCs that induce and prolong immunosuppressive endotypes. Aim 3. To identify the distinct immunosuppressive mechanisms of MDSCs from surgical sepsis patients over time, including immunometabolism, check-point inhibition, reactive oxygen and nitrogen production, and substrate availability. Using the established clinical infrastructure of the Sepsis and Critical Illness Research Center (SCIRC), a team science approach will be employed with collaborating PI's coming from multiple clinical and basic science disciplines. Aim 4. To test the hypothesis that in response to an initial inflammatory stimulus (severe blunt trauma) associated with a high risk of in-hospital sepsis, bone marrow (BM) hematopoietic stem cells (HSCs) promote immunosuppressive myelopoiesis at the expense of lymphopoiesis. With subsequent sepsis development, MDSCs induce their continued expansion through exocrine and paracrine signaling to HSCs. HSCs and MDSCs derived from severe blunt trauma patients will be analyzed for epigenetic and functional changes that initiate sepsis and continue the expansion of immunosuppressive MDSCs.

ELIGIBILITY:
Sepsis participant:

Inclusion Criteria:

1. age ≥18 years
2. meets criteria for sepsis/septic shock by Sepsis-3 consensus criteria.

Exclusion Criteria:

1. have disease states that predispose to significant immune system dysfunction
2. have comorbidity burden or goals of care that preclude recovery after sepsis. These criteria include:

   a. irreversible shock (death <12 hours) b. uncontrollable surgical source of sepsis c. patients deemed to be futile care or have advanced directives limiting resuscitative efforts d. alternative diagnoses causing shock state (e.g., hemorrhage, myocardial infarction or pulmonary embolus) e. known HIV infection with CD4+ count <200 cells/mm3 g. severe traumatic brain injury with unencumbered assessment of GCS equaling 3 on admission to the intensive care unit.
3. known pregnancy
4. enrollment >96 hours after suspected sepsis onset
5. pre-hospitalization bedridden performance status (WHO/Zubrod score ≥4)
6. subsequent clinical adjudication diagnosis not consistent with sepsis/septic shock by Sepsis-3 criteria.
7. Burn injury greater than 20% total body surface area (tBSA)

Trauma Participant:

Inclusion Criteria

1. All adults age ≥ 18 years
2. Blunt trauma patient with a. Injury Severity Score (ISS) greater than or equal to 25 b. ISS > 15 and one of the following: i. > 4 units of PRBC or >3 units of whole blood or >1500 ml of autogenous blood product in the first 24 hours of admission ii. AIS (acute injury score) > 2 spine iii. Shock on arrival (Systolic blood pressure (SBP) < 90)

OR

c. ISS > 15 and two of the following: i. Age > 55 ii. AIS > 2 chest iii. +ETOH (ethyl alcohol) on arrival iv. Any red blood cell transfusion in first 24 hours

Exclusion Criteria

1. Patients not expected to survive greater than 48 hours.
2. Prisoners.
3. Pregnancy.
4. Previous bone marrow transplantation.
5. Patients with End Stage Renal Disease.
6. Patients with any pre-existing hematological disease.
7. Patients deemed to be futile care or have advanced directives limiting resuscitative efforts.
8. Known HIV infection with CD4+ count <200 cells/mm3
9. Burn injury greater than 20% tBSA

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted to surgical and trauma intensive care units who screen positive for sepsis and are being treated by our standard-of-care sepsis protocol are candidates for the studies proposed in this proposal. For the purpose of these studies, sepsis will be defined using the new Sepsis-3 criteria.
  Patients admitted to the surgical and trauma intensive care units who have severe blunt trauma injury and have high risk of in-hospital sepsis.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
The total number of neutrophils and early myeloid derived suppressor cells will be measured and will be used to determine the magnitude of myelopoiesis dysfunction. | 6 months
  The total number of neutrophils and early Myeloid derived suppressor cells will be measured at sepsis onset and during hospitalization and at 3 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Lyle Moldawer, PhD, Principal Investigator — University of Florida; Philip Efron, MD, Principal Investigator — University of Florida; Tyler Loftus, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health at Shands hospital, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided